CLINICAL TRIAL: NCT05135533
Title: Cranial-nerve Non-invasive Neuromodulation and Dynamic Balance in Chronic Stroke Survivors
Brief Title: Neuromodulation and Dynamic Balance in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Brooks Rehabilitation (Other)
Responsible Party: Principal Investigator, Steven Kautz, Depertment Chair, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00113565
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Gait

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Portable Neuromodulation Stimulator (Experimental)
  Interventions: Device: Portable Neuromodulation Stimulation; Other: Gait and balance training
- Sham (Sham Comparator)
  Interventions: Device: Sham; Other: Gait and balance training

INTERVENTIONS:
Device: Portable Neuromodulation Stimulation — The PoNS group will receive electrical stimulation. Net direct current to the tongue electrode less than 1 µA (micro ampere) will be administered three times a week for four weeks in-lab setting, followed by three times a week for eight weeks at-home setting. Participants will continue to be enrolled in the study for additional 12 weeks without any intervention to evaluate long term effects.
  Arms: Portable Neuromodulation Stimulator
Device: Sham — The Sham group will not receive electrical stimulation.
  Arms: Sham
Other: Gait and balance training — During each session participants will receive gait training exercises for 20 minutes, 20 minutes of balance training exercises, and 20 minutes of breathing exercise three times a week for four weeks in-lab setting. This will be followed by 20 minutes of gait training exercises, 20 minutes of balance training exercises, and 20 minutes of breathing exercise three times a week for eight weeks at-home setting. Participants will continue to be enrolled in the study for additional 12 weeks without any intervention to evaluate long term effects.

SUMMARY:
Portable Neuromodulation Stimulator (PoNS) is non-invasive stimulation device placed on the tongue to stimulate those brain regions understood to be important for maintaining balance. This research study aims to collect evidence that PoNS therapy along with balance training improves postural and walking stability post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* At least six months since the onset of Ischemic or hemorrhagic stroke.
* Demonstrate residual paresis in the lower extremity (Fugl-Mayer lower extremity score < 34).
* Are able to provide informed consent demonstrated by their ability to weigh the consequences of participating versus not participating in the study.
* Can walk at least 10 feet with and without assistive device.
* Functional Gait Assessment score <22.

Exclusion Criteria:

* Pre-existing neurological disorders.
* Previous stroke affecting the other hemisphere .
* Severe arthritis or orthopedic problems that limit passive range of motion.
* Areas of recent bleeding or open wounds.
* Lack normal sensation on the tongue.
* Received treatment for cancer within the past year.
* Non-removable metal orthodontic devices.
* Oral health problems.
* Are sensitive to nickel, gold or copper.
* Chronic infectious diseases.
* Are pregnant.
* Have dementia

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | Pre-treatment, midpoint at four weeks, and post-treatment at 12 weeks
  Self-selected comfortable walking overground walking speed.
Change in balance | Pre-treatment, midpoint at four weeks, and post-treatment at at 12 weeks
  Functional Gait Assessment (FGA) assesses stability during walking. The score ranges between 0 and 30 with lower scores indicative of poor dynamic balance.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kautz, PhD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that underlie the results reported in the article, after de-identification.
Supporting Information: CSR
Time Frame: Immediately following publication no end date
Access Criteria: anyone who wishes to access the data